CLINICAL TRIAL: NCT03531398
Title: Postprandial Responses to Typical UK Meal Nutrient Profiles
Acronym: Pre-PREDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HR-17/18-5652
Record Dates: First submitted 2018-04-24; First posted 2018-05-21 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2018-04

CONDITIONS: Nutrition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fat meal (Experimental): Muffin containing 30g fat
  Interventions: Other: Metabolic test meal challenge
- Medium fat meal (Experimental): Muffin containing 20g fat
  Interventions: Other: Metabolic test meal challenge

INTERVENTIONS:
Other: Metabolic test meal challenge — Metabolic test meal challenge

SUMMARY:
The aim of the current study is to investigate the postprandial metabolic response to typically consumed fat and carbohydrate doses in single meals. An additional aim is to validate the use of dry blood spot (DBS) for triglyceride analysis versus venous blood sampling.

DETAILED DESCRIPTION:
Background: Dietary fat consumption is one of the major modifiable risk factors implicated in the causation of cardiovascular disease (CVD). Postprandial lipaemia (PPL); the increase in circulating blood triacylglycerol (TAG) concentrations after a fat containing meal, is an independent risk factor for cardiovascular disease. However, little is known about how different doses of fats as found in typical UK meals will influence the level of PPL.

The majority of research into PPL, including work by our own group and others has largely focused on the postprandial effect following high fat meals, with the primary goal of assessing mechanisms underlying fat metabolism. However, these findings are not relevant from a public health perspective; in reality the average fat content of a meal is much lower than this (~20- 30 g fat, (NDNS, 2013/4)); therefore it is important to assess the impact of doses of fat in this range on PPL to be relevant to public health. The few dose response studies that have been performed assessing fat load and PPL have used liquid test meals that are not relevant to every day meals.

PPL is usually measured by taking a series of blood samples from a cannula, however this is an invasive procedure. There has been an increase in the development of less invasive biochemical assessment, e.g. urine or saliva analysis or dried blood spot (DBS) analysis. DBS analysis is particularly advantageous as samples can be easily collected by the individual under assessment with minimal equipment and transferred easily for analysis via the post, providing simple home-testing. Frequently, postprandial research studies will draw blood from the cannula for multiple related outcomes and therefore, performing multiple assays from one DBS sample would be advantageous in minimizing participant discomfort.

Aim: The primary aim of the current study is to investigate the postprandial response following typical UK meal nutrient profiles containing 20-30g fat. Secondary aims will be to test the feasibility for measuring PPL, insulin, c-peptide and performing metabolomic analysis from DBS versus serum blood analysis. Further, it will assess the best practice for collection (venous versus finger prick) and storage (ambient versus freezer) of the DBS samples.

Hypothesis: Typical UK meal nutrient profiles will elicit detectable PPL. Further, DBS will be an effective method for measuring postprandial outcomes.

Expected value: The study will provide novel information on the effect of fat doses from typical UK meals on PPL. It will also provide feasibility for using DBS for measuring postprandial responses.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-65 years.
* Free of diagnosed diseases listed in exclusion criteria.
* Able to understand the information sheet and willing to comply with study protocol.
* Able to give informed consent.

Exclusion Criteria:

Refuse or are unable to give informed consent to participate in the study

* BMI >32 kg/m2
* BP >170/100 mm Hg
* Have had long term inflammatory disease or cancer in the last three years.
* Have had long term gastrointestinal disorders including inflammatory bowel disease (IBD) or Coeliac disease (gluten allergy).
* Are taking the following daily medications: immunosuppressants, antibiotics in the last three months
* Are long-term users of PPIs, unless they are able to stop two weeks before the start of the study.
* Have type I diabetes mellitus or type II diabetes mellitus.
* Are currently suffering from acute clinically diagnosed depression.
* Have had a heart attack (myocardial infarction) or stroke in the last 6 months.
* Are pregnant
* Are vegan, suffering from an eating disorder or unwilling to take foods that are part of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self identification from a questionnaire if male or female
Enrollment: 17 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Postprandial lipaemia | 0-4 hours postprandially
  Change in serum triglycerides

SECONDARY OUTCOMES:
Postprandial glycaemia | 0-4 hours postprandially
  Change in plasma glucose

OTHER OUTCOMES:
Postprandial plasma insulin | 0-4 hours postprandially
  Change in plasma insulin
Postprandial plasma c-peptide | 0-4 hours postprandially
  Change in plasma C-peptide

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Berry, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No